CLINICAL TRIAL: NCT05504408
Title: A Retrospective and Prospective Multicenter Observational Study for the Evaluation of Incidence of Systemic Mastocytosis With Associated t(8;21) Acute Myeloid Leukemia in t(8;21) Acute Myeloid Leukemia
Brief Title: Observational Study for the Evaluation of Incidence of Systemic Mastocytosis in t(8;21) Acute Myeloid Leukemia
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: The First Affiliated Hospital of Soochow University (Other)
Responsible Party: Principal Investigator, Chen Suning, Director, Clinical Professor, The First Affiliated Hospital of Soochow University
Other Study IDs: SM-AML01
Record Dates: First submitted 2022-08-04; First posted 2022-08-17 (Actual); Last update posted 2023-10-10 (Actual); Status verified 2023-10

CONDITIONS: Systemic Mastocytosis With AHNMD; Acute Myeloid Leukemia With T(8;21)(Q22;Q22)

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 24 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Systemic Mastocytosis with associated t(8;21) AML: SM and AML were diagnosed according to the 5th edition WHO classification criteria.
- The t(8;21) AML without Systemic Mastocytosis: The t(8;21) AML patients do not have associated Systemic Mastocytosis according to the 5th edition WHO classification criteria and no AML1-ETO clone was detected in mast cells.
- OSM (Oligo-mastocytic SM) with associated t(8;21) AML: The t(8;21) AML patients do not have associated Systemic Mastocytosis according to the 5th edition WHO classification criteria, but AML1-ETO clones were detected in mast cells.

SUMMARY:
The observational study aimed at evaluating the incidence of systemic mastocytosis associated with t(8;21) AML in patients with de novo t(8;21) AML and their responses to first induction, and the prognosis from standard therapy.

DETAILED DESCRIPTION:
This is a multicenter, retrospective and prospective, observational study that aims to collect clinical information on patients with systemic mastocytosis associated with t(8;21) AML from September 2022 to August 2023. No intervention is expected.

The purpose of this study is to identify and characterize the patients with systemic mastocytosis associated with t(8;21) AML, t(8;21) AML without systemic mastocytosis, and OSM (Oligo-mastocytic SM) with associated t(8;21) AML.

In order to estimate the incidence of systemic mastocytosis associated with t(8;21) AML, a survey will be sent every month to all participating sites to collect the number of all diagnoses of systemic mastocytosis associated with t(8;21) AML, t(8;21) AML without systemic mastocytosis, and OSM with associated t(8;21) AML. All patients will be followed until August 2025 in order to have at least 2 years of observation.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, Age (years) >= 5;
2. Newly diagnosed as t(8;21) AML patients according to World Health Organization (WHO) classification;
3. Patients who sign the informed consent must have the ability to understand and be willing to participate in the study and sign the informed consent.

Exclusion Criteria:

1. The t(8;21) AML patients with SM have been diagnosed already;
2. Patients with drug abuse or long-term alcoholism that affected the evaluation of trial results;
3. Patients were deemed unsuitable for enrolment by the investigator.

Min Age: 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Candidates will come from patients with newly diagnosed t(8;21) acute myeloid leukemia (AML) in the First Affiliated Hospital of Soochow University and the participated centers from September 2022.
  Participants should meet the inclusion criteria and not meet exclusion criteria.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2022-09-01 (Actual); Primary Completion 2024-08-31 (Estimated); Study Completion 2024-08-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of Systemic Mastocytosis associated with t(8;21) Acute Myeloid Leukemia | at 1 year
  Evaluation of the incidence of systemic mastocytosis associated with t(8;21) AML in patients with de novo t(8;21) AML.
  The incidence of systemic mastocytosis associated with t(8;21) AML will be evaluated by means of the number of diagnosis of systemic mastocytosis associated with t(8;21) AML on the number of all diagnoses of de novo t(8;21) AML between September 2022 and August 2023.

SECONDARY OUTCOMES:
Hematological characteristics of all the t(8;21) Acute Myeloid Leukemia | at 1 year
  1. The neutrophils, eosinophils, basophils, and mast cells in WBC classification (%);
  2. The proliferative degree in sections of BM (%);
  3. The ratio of mast cells in BM smear and FCM (%);
  4. The ratio of expression of CD25, CD2, and CD30 in FCM (%);
  5. The quantification of the AML1-ETO gene fusions (%).
Responses to the first induction therapy of all the t(8;21) Acute Myeloid Leukemia | at 1 year
  1. The rate of eligible complete remission (CR) patients(%);
  2. The rate of eligible CR with incomplete hematologic recovery (CRi) patients(%);
  3. The rate of eligible morphologic leukemia-free state (MLFS) patients(%);
  4. The rate of eligible partial remission (PR) patients(%);
  5. The rate of eligible no response (NR) patients(%);
  6. The rate of eligible CR without MRD patients(%);
  7. The rate of eligible overall response rate (ORR) patients(%).
Incidence of transplantation of all the t(8;21) Acute Myeloid Leukemia | at 1 year
  The outcome of transplant in three groups of patients with systemic mastocytosis associated with t(8;21) AML, t(8;21) AML without systemic mastocytosis, and OSM with associated t(8;21) AML.
Survival Distribution of all the t(8;21) Acute Myeloid Leukemia | at 2 years
  1. Overall survival (months): Measured the time from enrollment to the date of the last follow-up or death;
  2. Leukemia-free survival (months): Measured the time from the date of attaining CR1 until the first relapse, death, or the final follow-up day.

CONTACTS AND LOCATIONS:
Overall Officials: Suning Chen, professor, Principal Investigator — The First Affiliated Hospital of Soochow University, Jiangsu Institute of Hematology
Locations (1):
- The First Affiliated Hospital of Soochow University, Jiangsu Institute of Hematology, Suzhou, Jiangsu, China